CLINICAL TRIAL: NCT04288388
Title: The Effect Of Ice Massage Applied To The Hand During Episiotomy Repair On Perceived Pain
Brief Title: The Effect Of Ice Massage On Perceıved Pain
Acronym: icemassage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Bihter Akın, Asisstant Prof. Dr., Selcuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Ice Massage
Record Dates: First submitted 2020-02-07; First posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Labor Pain; Episiotomy Wound
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Intervention Model Description: The study group being 178 and the control group being 169 with 347 women. Immediately before the episiotomy repair was started (after exit of placenta and applying local anesthetic agent), women assigned to the study (massage) group were asked to place plastic gloves filled with ice pieces in the LI4 point on hand. This application was made for 5 minutes to the right hand and for 5 minutes to the left hand. Women were asked to mark the perceived pain level before the application and at the end of the application using the VAS (Visual Analog Scale) (perceived pain level during episiotomy repair). In the control group women were not excluded from routine practice; women were asked to mark the perceived pain level before episiotomy repair begin and at the end the repair using the VAS (Visual Analog Scale) (perceived pain level during episiotomy repair) like the study (massage) group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- massage group (Experimental): Immediately before the episiotomy repair was started (after exit of placenta and applying local anesthetic agent), women assigned to the study (massage) group were asked to place plastic gloves filled with ice pieces in the LI4 point on hand. This application was made for 5 minutes to the right hand and for 5 minutes to the left hand. The episiotomy was opened by the same midwife as all the women to the right mediolateral and repaired by the same midwife with the same technique and material.The ice massage was repeated until the episiotomy repair was over; total massage time and episiotomy repair time were recorded. Women were asked to mark the perceived pain level before the application and at the end of the application using the VAS (Visual Analog Scale) (perceived pain level during episiotomy repair).
  Interventions: Behavioral: massage group
- Control group (No Intervention): I the control group women were not excluded from routine practice; women were asked to mark the perceived pain level before episiotomy repair begin and at the end the repair using the VAS (Visual Analog Scale) (perceived pain level during episiotomy repair) like the study (massage) group.

INTERVENTIONS:
Behavioral: massage group — In recent years, in the literature, it is known that many non-pharmacological techniques are applied to reduce the pain of birth in addition to local anesthesia. One of these nonpharmacological methods is the application of pressure to LI4 point on hand with ice.
  Other Names: ice massage
  Arms: massage group

SUMMARY:
Introduction: In this study, it was aimed to examine the effect of ice massage applied to the hand during episiotomy repair on perceived pain.

Methods: The study was carried out in the delivery unit of a maternity hospital between April 15, 2018 and November 15, 2018 with vaginal delivery for the first time, no complication developed during the delivery, with the study group being 178 and the control group being 169 with 347 women. Immediately before the episiotomy repair was started (after exit of placenta and applying local anesthetic agent), women assigned to the study (massage) group were asked to place plastic gloves filled with ice pieces in the LI4 point on hand. This application was made for 5 minutes to the right hand and for 5 minutes to the left hand. The episiotomy was opened by the same midwife as all the women to the right mediolateral and repaired by the same midwife with the same technique and material.The ice massage was repeated until the episiotomy repair was over; total massage time and episiotomy repair time were recorded. Women were asked to mark the perceived pain level before the application and at the end of the application using the VAS (Visual Analog Scale) (perceived pain level during episiotomy repair). In the control group women were not excluded from routine practice; women were asked to mark the perceived pain level before episiotomy repair begin and at the end the repair using the VAS (Visual Analog Scale) (perceived pain level during episiotomy repair) like the study (massage) group. Data were evaluated by using chi square, student t test and ANOVA in SPSS 18.0 program. In order to carry out this study , the necessary consent was obtained from the ethics committee, institution and women.

DETAILED DESCRIPTION:
Introduction: Episiotomy is the most common surgical intervention during vaginal delivery. Perineal damage during this incision causes perineal pain; pain and anxiety levels of women increase during episiotomy repair as well as during labor and delivery. In order to minimize this level of pain, local anesthetic agents are routinely administered to the episiotomy region. In recent years, in the literature, it is known that many non-pharmacological techniques are applied to reduce the pain of birth in addition to local anesthesia. One of these nonpharmacological methods is the application of pressure to LI4 point on hand with ice. Although there are studies conducted to reduce the pain with LI4 point in the literature, the studies done to reduce the pain experienced during episiotomy repair are quite limited.In this study, it was aimed to examine the effect of ice massage applied to the hand during episiotomy repair on perceived pain.

Methods: The study was carried out in the delivery unit of a maternity hospital between April 15, 2018 and November 15, 2018 with vaginal delivery for the first time, no complication developed during the delivery, with the study group being 45 and the control group being 60 with 105 women. Immediately before the episiotomy repair was started (after exit of placenta and applying local anesthetic agent), women assigned to the study (massage) group were asked to place plastic gloves filled with ice pieces in the LI4 point on hand. This application was made for 5 minutes to the right hand and for 5 minutes to the left hand. The episiotomy was opened by the same midwife as all the women to the right mediolateral and repaired by the same midwife with the same technique and material.The ice massage was repeated until the episiotomy repair was over; total massage time and episiotomy repair time were recorded. Women were asked to mark the perceived pain level before the application and at the end of the application using the VAS (Visual Analog Scale) (perceived pain level during episiotomy repair). In the control group women were not excluded from routine practice; women were asked to mark the perceived pain level before episiotomy repair begin and at the end the repair using the VAS (Visual Analog Scale) (perceived pain level during episiotomy repair) like the study (massage) group. Data were evaluated by using chi square, student t test and ANOVA in SPSS 18.0 program.

ELIGIBILITY:
Inclusion Criteria:

18-40 years having a vaginal birth with episiotomy

Exclusion Criteria:

Under 18 years (adolesant women)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 347 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Vas | ten minute after ice massage
  A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms.Using a ruler, the score is determined by mea-suring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity. Based on the distribution of pain VAS scores in post- surgical patients (knee replacement, hyster-ectomy, or laparoscopic myomectomy) who described their postoperative pain intensity as none, mild, moderate, or severe, the following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm)

CONTACTS AND LOCATIONS:
Overall Officials: Birsen Karaca Saydam, PhD, Study Director — Ege University
Locations (1):
- Selcuk University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No